CLINICAL TRIAL: NCT00034671
Title: Phase II Study of Safety, Tolerance, Efficacy, and Pharmacokinetics of Posaconazole (SCH 56592) for the Treatment of Invasive Fungal Infections in Immunocompromised Hosts
Brief Title: PK/PD Study of Posaconazole for Empiric Treatment of Invasive Fungal Infections in Neutropenic Patients or Treatment of Refractory Invasive Fungal Infections (Study P01893)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01893
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Mycoses
Keywords: Aspergillosis, Candidiasis, Mucormycosis, Cryptococcosis; Invasive Fungal Infections
MeSH Terms: conditions — Mycoses; Aspergillosis; Candidiasis; Mucormycosis; Cryptococcosis; Invasive Fungal Infections

INTERVENTIONS:
Drug: Posaconazole oral suspension

SUMMARY:
This phase II study will be conducted to:

1. evaluate the pharmacokinetics, safety, tolerance, and efficacy of different dosing schedules of Posaconazole in immunocompromised hosts with a variety of refractory invasive fungal infections or in subjects who require empiric antifungal therapy and
2. identify the dosing schedule that provides the most consistent therapeutic drug exposure in this patient population.

DETAILED DESCRIPTION:
This is an open-label, randomized, parallel group, study of pharmacokinetics, safety, tolerance, and efficacy of Posaconazole in the treatment of immunocompromised hosts with refractory invasive fungal infections or in subjects who require empiric antifungal therapy.

The projected number of subjects planned for enrollment is 100 evaluable subjects. The number of planned study sites is approximately ten in the United States and approximately eight in the rest of the world.

ELIGIBILITY:
Inclusion Criteria:

* A proven, either probable or possible invasive fungal infection which is refractory to standard antifungal therapies.
* Subjects who received >72 hours of systemic empiric antibacterial therapy and are neutropenic (<500 neutrophils per mm3 and, have had fever that has reached an oral temperature >38c (or >100.4f)twice in the last 48 hours, or

have a recurrence of fever (oral temperature, >38c or >100.4F) while receiving broad spectrum antibacterial therapy after prior resolution of fever while on antibacterial therapy.

* Able to take oral medication or take medication via enteral feeding tube.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2001-01; Primary Completion 2001-11 (Actual); Study Completion 2002-03 (Actual)

REFERENCES:
- [Result] Ullmann AJ, Cornely OA, Burchardt A, Hachem R, Kontoyiannis DP, Topelt K, Courtney R, Wexler D, Krishna G, Martinho M, Corcoran G, Raad I. Pharmacokinetics, safety, and efficacy of posaconazole in patients with persistent febrile neutropenia or refractory invasive fungal infection. Antimicrob Agents Chemother. 2006 Feb;50(2):658-66. doi: 10.1128/AAC.50.2.658-666.2006. PMID 16436724